CLINICAL TRIAL: NCT02464046
Title: A Randomized, Placebo-controlled, 2-way Crossover, Double-blind Study to Evaluate the Efficacy, Safety and Tolerability of JNJ-42847922 in Subjects With Insomnia Disorder Without Psychiatric Comorbidity
Brief Title: Study to Evaluate Efficacy, Safety and Tolerability of JNJ-42847922 in Participants With Insomnia Disorder Without Psychiatric Comorbidity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR107585; 42847922ISM2002 (Other: Janssen Research & Development, LLC); 2015-001672-22 (EudraCT Number)
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Insomnia
Keywords: Insomnia; JNJ-42847922; Placebo
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- JNJ-42847922 then Placebo (Experimental): Participants receive 2*20 milligram (mg) tablet of JNJ-42847922 orally once daily from Day 1 to Day 5 of period 1. After a washout period of 5 to 9 days participants will receive matching placebo from Day 1 to Day 5 of period 2.
  Interventions: Drug: JNJ-42847922; Drug: Placebo
- Placebo then JNJ-42847922 (Experimental): Participants will receive matching placebo from Day 1 to Day 5 of period 1. After a washout period of 5 to 9 days participants will receive 2*20 mg tablet of JNJ-42847922 orally once daily from Day 1 to Day 5 of period 2.
  Interventions: Drug: JNJ-42847922; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42847922 — Participants in arm JNJ-42847922 then Placebo will receive 2*20 mg tablet of JNJ-42847922 orally once daily from Day 1 to Day 5 in Period 1 and participants in arm Placebo then JNJ-42847922 will receive 2*20 mg tablet of JNJ-42847922 orally once daily from Day 1 to Day 5 in Period 2.
Drug: Placebo — Participants in arm JNJ-42847922 then Placebo will receive matching Placebo orally once daily from Day 1 to Day 5 in Period 2 and participants in arm Placebo then JNJ-42847922 will receive matching placebo orally once daily from Day 1 to Day 5 in Period 1.

SUMMARY:
The primary purpose of this study is to investigate the effect of JNJ-42847922 (change versus placebo) on sleep efficiency (SE) measured by polysomnography (PSG) after single and multiple dose administration to participants with insomnia disorder without psychiatric comorbidity.

DETAILED DESCRIPTION:
This is a multi-center, randomized (study medication assigned to participants by chance), placebo-controlled, double-blind (neither physician nor participant knows the identity of the assigned treatment), 2-way cross-over study of JNJ-42847922 participants with insomnia disorder without psychiatric comorbidity. The study consists of following phases: screening (28 days prior to Day 1), a double-blind treatment phase (consists of 5-day treatments, either JNJ-42847922 or placebo in subsequent 2-treatment periods, each separated with washout period of 5 to 9 days), and a follow-up examination (7 to 14 days after last dose administration). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants aged between 18 and 65 years, inclusive
* Body mass index (BMI) between 18 and 30 kilogram per square meters (kg/m^2) inclusive (BMI = weight/height^2)
* Insomnia Severity Index (ISI) score more than or equal to (>=) 15 at screening
* Insomnia: at screening participants will report both difficulties with sleep onset and sleep maintenance. Insomnia will furthermore objectively be established prior to enrollment per PSG recorded over 3 consecutive nights. Participants will sleep for 3 consecutive nights in the sleep center. First and second night data will be used to exclude any participant with restless leg syndrome, apnea, parasomnias or other sleep disorders. On the second and third night participants are required to meet objective inclusion criteria: 2-night mean LPS of >=30 minutes with no night <20 minutes, and on both nights TST <=6 hours and wake after sleep onset (WASO) >30 minutes
* Participants must be healthy / medically stable on the basis of clinical laboratory tests, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and baseline

Exclusion Criteria:

* Participant has current signs/symptoms of, liver or renal insufficiency; hypothyroidism or hyperthyroidism, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, or metabolic disturbances. Participants with non-insulin dependent diabetes mellitus who are adequately controlled (not on insulin) may participate in the study
* History of epilepsy or fits or unexplained black-outs
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or admission
* Clinically significant abnormal physical and neurological examination, vital signs or 12-lead ECG at screening or baseline
* Smoking >=10 cigarettes/daily
* Insomnia related to restless leg syndrome, sleep breathing disorder, narcolepsy, obstructive sleep apnea/hypopnea, central sleep apnea, sleep-related hypoventilation, circadian rhythm sleep-wake disorders, substance/medication-induced sleep disorder or parasomnias
* Night-shift worker or significantly shifted diurnal activity pattern

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency by Polysomnography | up to Night 5
  The total sleep time divided by the total time in bed (that is, the number of minutes from the beginning of the Polysomnography recording to the end of the recording).

SECONDARY OUTCOMES:
Total Sleep Time by Polysomnography | up to Night 5
  All of the minutes of Stages 1, 2, 3/4 Non Rapid Eye-Movement (NREM) and Rapid-Eye-Movement (REM) sleep, as measured by Polysomnography, are summed to determine the Total Sleep Time.
Wake Time After Sleep Onset by Polysomnography | up to Night 5
  The number of minutes in the Awake stage after the onset of persistent sleep to the end of the recording.
Number of Awakenings After Persistent Sleep by Polysomnography | up to Night 5
  Number of Awakenings is defined as the number of times after the onset of persistent sleep that there is a wake entry of at least 2 epochs in duration. Each entry must be separated by Stage 2, 3/4 NREM sleep or REM sleep in order to be counted.
Total Time Spent in Deep Sleep by Polysomnography | up to Night 5
  Duration of slow wave sleep will be reported.
Mean Latency to Persistent Sleep by Polysomnography | up to Night 5
  Elapsed time from the beginning of the Polysomnography recording to the onset of the first 10 minutes of continuous sleep will be measured over 2 nights and the average time to sleep will be calculated.
Leeds Sleep Evaluation Questionnaire (LSEQ) Score | up to Night 5
  The LSEQ is a participant-reported 10-item visual analogue scale score used to rate the quality of sleep and to assess changes in sleep quality over the course of treatment.
Subjective assessment of sleep by Questionnaire | up to Night 5
  Subjective assessment of sleep parameters will be assessed by following questions to indicate how much and how well participant slept during the past night: 1. How long did it take you to fall asleep for the first time (Mean Subjective sleep onset latency); 2. How long have you slept in total (Total sleep time); 3. How long were you awake after initial sleep onset until you finally got out of bed (Wake After Sleep Onset); 4. How often did you awake during the night (how many times); 5. How did you rate the quality of the night sleep (1= extremely bad 10 =excellent).
Next Morning Residual Effects by Bond and Lader Visual Analogue Scale | up to Night 5
  The Bond and Lader Visual Analogue Scale consists of sixteen 100 mm visual analog scales anchored by antonyms (example, Alert-Drowsy, Lethargic-Energetic, etc). Scores will be combined to form three mood factors: alertness, calmness, and contentedness.
Next Morning Residual Effects by cognitive test battery | up to Night 5
Next Morning Residual Effects by Karolinska Sleepiness Scale | up to Night 5
  The KSS is a participant-reported assessment used to rate sleepiness on a scale of 1 to 9, ranging from 'extremely alert' (1) to 'very sleepy, great effort to keep awake, fighting sleep (9).
Number of Participants with Adverse Events (AEs) and Serious AEs | up to Night 5
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- Hollywood, Florida, United States
- Germany (3):
  - Berlin
  - Hamburg
  - Schwerin
- Leiden, Netherlands

REFERENCES:
- [Derived] De Boer P, Drevets WC, Rofael H, van der Ark P, Kent JM, Kezic I, Parapatics S, Dorffner G, van Gerven J, Benes H, Keicher C, Jahn H, Seiden DJ, Luthringer R. A randomized Phase 2 study to evaluate the orexin-2 receptor antagonist seltorexant in individuals with insomnia without psychiatric comorbidity. J Psychopharmacol. 2018 Jun;32(6):668-677. doi: 10.1177/0269881118773745. Epub 2018 May 31. PMID 29848147